CLINICAL TRIAL: NCT03647150
Title: Treatment of High-Risk Moderate Acute Malnutrition Using Expanded Admission Criteria (Hi-MAM Study): A Cluster-randomized Controlled Trial Protocol
Brief Title: Treatment of High-Risk Moderate Acute Malnutrition Using Expanded Admission Criteria
Acronym: Hi-MAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Centre for Global Child Health, Hospital for Sick Kids, Toronto, Canada (Unknown); Department of Psychology, University of Tampere, Finland (Unknown); Project Peanut Butter, Sierra Leone (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201807153
Record Dates: First submitted 2018-07-31; First posted 2018-08-27 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Acute Malnutrition (MAM) (Other): MAM children at control clinics or MAM children at intervention clinics that do no have high rick characteristics. Control treatment is "Mother Care" counselling, delivered by a respected elder in the local community.
  Interventions: Behavioral: Mother Care group
- High Risk Moderate Acute Malnutrition (MAM) (Experimental): The intervention treatment incorporates Mother Care counselling, provision of one packet (508 calories) of ready-to-use therapeutic food (RUTF) daily and a 1 week course of amoxicillin. This provision will continue until the child has reached a mid-upper arm circumference (MUAC) equal to or greater than 12.5 cm or 12 weeks have elapsed.
  Interventions: Drug: amoxicillin; Dietary Supplement: Ready-to-use therapeutic food (RUTF); Behavioral: Mother Care group

INTERVENTIONS:
Drug: amoxicillin — At enrollment the child will receive a 1 week course of amoxicillin
  Arms: High Risk Moderate Acute Malnutrition (MAM)
Dietary Supplement: Ready-to-use therapeutic food (RUTF) — 1 sachet RUTF per day (508 calories) till child MUAC is greater than 12.4 cm or 12 weeks have elapsed
  Arms: High Risk Moderate Acute Malnutrition (MAM)
Behavioral: Mother Care group — Nutrition education via mother care groups lead by a respected elder in the local community

SUMMARY:
This project explores whether children have better growth and cognitive development when the clinic identifies "higher risk" MAM children and support them either with the same treatment as SAM children or with the recommended practice: nutrition counseling.

DETAILED DESCRIPTION:
This is a cluster-randomized controlled trial taking place in 20 community clinics providing malnutrition care in Sierra Leone.

All participants will be children aged 6-59 months. Control participants will have moderate acute malnutrition (MAM), defined as mid-upper arm circumference (MUAC) 11.5-<12.5. High Risk MAM will be defined with a MUAC 11.5 to <11.9 or WAZ<-3.5 or Mother not the caretaker or not breastfeeding at <2 years old. Low risk MAM defined with a MUAC 11.9 to <12.5 with no risk factors.

Control group and low risk group caregiver's will received nutrition education via mother care groups every two weeks for 6 weeks and will be followed up 12 and 24 weeks post-enrollment.

High risk group will receive 1 week supply of amoxicillin at enrollment and 1 sachet of RUTF per day till MUAC is equal to or greater than 12.5 or up to 12 weeks of treatment. Their caregiver will also receive nutrition education via the mother care groups. The investigators will also follow up with the participant at 12 and 24 weeks post-enrollment.

A subset of the participants in each group will also be enrolled in a cognitive development substudy were the investigators will be using a eye tracking performance assessment. Investigators will also enroll health adult participants for eye tracking assessment. Adult data will be used as a reference when interpreting results.

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated MAM (based on MUAC equal to or greater than 11.5 cm and <12.5)

Exclusion Criteria:

* currently involved in another research trial or feeding program
* medical complication such as oedema, severe nausea/vomiting, severe dehydration, or severe pneumonia
* have a diagnosed or visible sign of developmental delay
* have a history of peanut or milk allergy

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1322 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Recovery from moderate acute malnutrition (MAM) | up to 12 weeks of treatment
  proportion of participants recovered based on mid-upper arm circumference(MUAC) Recovery is defined as MUAC greater than or equal to 12.5cm before or at 12 weeks after enrollment.

SECONDARY OUTCOMES:
Participant survival rates | Duration of the study 24 weeks post-enrollment
  Proportion of participants survival rates during the study
Participants deterioration to severe acute malnutrition(SAM) | Duration of the study 24 weeks post-enrollment
  Proportion of participants that deteriorate from moderate acute malnutrition(MAM) to severe acute malnutrition(SAM). SAM is defined at mid-upper arm circumference(MUAC)<11.5 or presence of oedema.
Participants that remain or become underweight using weight for age z-score | 24 weeks post-enrollment
  the difference between the weight for age z-score(WAZ) from enrollment to 24 weeks post-enrollment
Participants that remain or become Stunted | 24 weeks post-enrollment
  the difference between length for age z-score(LAZ) from enrollment to 24 weeks post enrollment
Participants that remain or become Wasted | 24 weeks post-enrollment
  the difference between weight for length z-score(WHL) from enrollment to 24 weeks post enrollment
Eye tracking performance for cognitive development | 24 weeks post enrollment
  the difference between the eye tracking performance from enrollment to 24 weeks post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Mark Manary, MD, Principal Investigator — Washington University School of Medicine in St. Louis
Locations (1):
- Project Peanut Butter, Freetown, Sierra Leone

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joshua GE, Jadhav M, Bhaktaviziam A, Mokashi S. Mental retardation in children. II. Leucodystrophies. Indian Pediatr. 1974 Jan;11(1):53-9. No abstract available. PMID 4839581
- [Background] Lenters LM, Wazny K, Webb P, Ahmed T, Bhutta ZA. Treatment of severe and moderate acute malnutrition in low- and middle-income settings: a systematic review, meta-analysis and Delphi process. BMC Public Health. 2013;13 Suppl 3(Suppl 3):S23. doi: 10.1186/1471-2458-13-S3-S23. Epub 2013 Sep 17. PMID 24564235
- [Background] Chang CY, Trehan I, Wang RJ, Thakwalakwa C, Maleta K, Deitchler M, Manary MJ. Children successfully treated for moderate acute malnutrition remain at risk for malnutrition and death in the subsequent year after recovery. J Nutr. 2013 Feb;143(2):215-20. doi: 10.3945/jn.112.168047. Epub 2012 Dec 19. PMID 23256140
- [Background] Maust A, Koroma AS, Abla C, Molokwu N, Ryan KN, Singh L, Manary MJ. Severe and Moderate Acute Malnutrition Can Be Successfully Managed with an Integrated Protocol in Sierra Leone. J Nutr. 2015 Nov;145(11):2604-9. doi: 10.3945/jn.115.214957. Epub 2015 Sep 30. PMID 26423737
- [Background] Ekelund U, Ong KK, Linne Y, Neovius M, Brage S, Dunger DB, Wareham NJ, Rossner S. Association of weight gain in infancy and early childhood with metabolic risk in young adults. J Clin Endocrinol Metab. 2007 Jan;92(1):98-103. doi: 10.1210/jc.2006-1071. Epub 2006 Oct 10. PMID 17032722
- [Background] Khara T, Mwangome M, Ngari M, Dolan C. Children concurrently wasted and stunted: A meta-analysis of prevalence data of children 6-59 months from 84 countries. Matern Child Nutr. 2018 Apr;14(2):e12516. doi: 10.1111/mcn.12516. Epub 2017 Sep 25. PMID 28944990
- [Background] Schofield C, Ashworth A. Why have mortality rates for severe malnutrition remained so high? Bull World Health Organ. 1996;74(2):223-9. PMID 8706239
- [Derived] Lelijveld N, Godbout C, Krietemeyer D, Los A, Wegner D, Hendrixson DT, Bandsma R, Koroma A, Manary M. Treating high-risk moderate acute malnutrition using therapeutic food compared with nutrition counseling (Hi-MAM Study): a cluster-randomized controlled trial. Am J Clin Nutr. 2021 Sep 1;114(3):955-964. doi: 10.1093/ajcn/nqab137. PMID 33963734
- See also: United Nations Department of Economic and Social Affairs, P.D. World Population Prospectus 2017. 2017 — https://esa.un.org/unpd/wpp/DataQuery/
- See also: WHO. IMCI chart booklet. 2014 — http://www.who.int/maternal_child_adolescent/documents/IMCI_chartbooklet/en/